CLINICAL TRIAL: NCT03192423
Title: Acute Mental Stress Among the Physician and Patient During Lumbar Puncture, and Its Impact on Performance and Patient Related Outcomes
Brief Title: Acute Mental Stress During Lumbar Puncture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Region Zealand (Other)
Responsible Party: Principal Investigator, Mikael Johannes Vuokko Henriksen, Principal Investigator, MD, Rigshospitalet, Denmark
Other Study IDs: AMSLP
Record Dates: First submitted 2017-06-13; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Stress, Emotional; Spinal; Puncture, Complications, Headache; Lumbar Puncture
Keywords: Stress; Performance of procedures; Lumbar Puncture
MeSH Terms: conditions — Stress, Psychological; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Expert: The physicians in the Expert-group will perform a LP following local standard procedure protocol.
- Intermediate: The physicians in the Intermediate-group will perform a LP following local standard procedure protocol.
- Novice: The physicians in the novice-group will perform a LP following local standard procedure protocol.

SUMMARY:
This study explores lumbar puncture operators stress associated with their performance of the procedure, across three experience levels: Experts, Intermediates, and Novices.

The study will investigate the association of this potential stress to patient experienced stress and patient related outcomes of the lumbar puncture procedure.

DETAILED DESCRIPTION:
The consequences of being in a state of Acute Mental Stress are reduced working memory, decreased psychomotor performance, and impaired performance. Although some levels of increased stress response might be beneficial, there seems to be an upper-limit when performance is reduced.

According to the Cognitive Activation Theory of Stress (CATS), the stress sensation arises when the requirements exceed the resources for a given task. For the LP procedure, a stress sensation among novice residents might arise due to the combination of the LP being a complex procedure depending on both technical as non-technical aspects combined with residents uncertainties for procedural performance and a fear of doing harm.

Despite a growing recognition of stress among residents, the acute mental stress of residents performing invasive procedures has been unacknowledged. Within neurology, internal medicine, and emergency medicine a particular subject for this stress might pertain to residents' first performance of the lumbar puncture.

However, for non-surgical invasive procedures as the LP, there is a lack of evidence for measurements of AMS across experience levels and how this potential stress might influence the performance and patient related outcomes.

Hence, the aim of this study is to explore stress levels across lumbar puncture experience levels and how this potential stress might affect procedural performance and the patients' experience of stress and outcomes of the procedure. Additionally, the study will explore a potential correlation between patient stress and the risk of developing post-dural puncture headache.

ELIGIBILITY:
Physicians:

Inclusion Criteria physicians:

* Medical Doctor or Medical student working as substitute junior medical officer
* Speaking Danish fluently
* Understanding and accepting study implications
* For novice group only: Medical student having clinical rotation at the study sites

Exclusion Criteria physicians:

* N/A

For expert group physicians: Consultant (or other senior physician position); LP experience > 100 procedures; supervisor for novice performer; Performing LP on a regular basis.

For intermediate group physicians:

Performing LP on a regular basis; LP experience of 10-80 procedures.

For novice group physicians:

No previous lumbar puncture experience

For patients enrolled in the study:

Inclusion Criteria Patients:

* Referred to the outpatient clinic for a LP;
* Glasgow Coma Scale 15;
* Proficiency in the Danish Language;
* Age between 18 and 80 years;
* Understanding and accepting study implications
* Able to co-operate to the procedure without a need for personal assistance;
* Providing written and orally informed consent

Exclusion Criteria Patients:

* Lumbar puncture intended on suspicion of Alzheimer or another dementia diagnosis;
* Cognitive impairment, assessed by the study investigator or local nurse/doctor; -
* Physical disabilities, requiring personal assistance.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Physicians:
  Physicians working at departments with frequent performance of LP. Physicians should represent the three experience levels novices, intermediates and experts.
  Patients:
  All patients referred for a lumbar puncture with respect to inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-07-01 (Estimated); Study Completion 2017-08-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Appraisal | Five minutes before performance
  Cognitive Appraisal explores the individuals perception of resources and demands for the performance (scores range from 1/6 to 6)
State Trait Anxiety Inventory - Short (before performance) | Five minutes before performance
  A questionaire exploring the stress related anxiety
State Trait Anxiety Inventory - Short (during performance) | Just before needle insertion
  A questionaire exploring the stress related anxiety
Heart Rate Variability before performance (Heart rate) | A recording of 5 minutes obtained five minutes before performance.
  Heart Rate Variability: Heart rate (bp/min)
Heart Rate Variability before performance (Spectrum analysis) | A recording of 5 minutes obtained five minutes before performance.
  Heart Rate Variability: Total power (Sum of Low Frequency, Very Low frequency, High Frequency) (ms)
Heart Rate Variability before performance (Spectrum analysis) | A recording of 5 minutes obtained five minutes before performance.
  Heart Rate Variability: LF/HF - ratio
Heart Rate Variability before performance (Timedomain analysis) | A recording of 5 minutes obtained five minutes before performance.
  Heart Rate Variability before performance Timedomain analysis: RMSDD (ms), pNN50 (%)
Heart Rate Variability during performance (Heart rate) | A recording of 5 minutes obtained five minutes before obtaining liquor or abandoning the procedure.
  Heart Rate Variability: Heart rate (bp/min)
Heart Rate Variability during performance (Spectrum analysis) | A recording of 5 minutes obtained five minutes before obtaining liquor or abandoning the procedure.
  Heart Rate Variability: Total Power (Sum of Low Frequency, Very Low frequency, High Frequency) (ms)
Heart Rate Variability during performance (Spectrum analysis) | A recording of 5 minutes obtained five minutes before obtaining liquor or abandoning the procedure.
  Heart Rate Variability: LF/HF - ratio
Heart Rate Variability during performance (Timedomain analysis) | A recording of 5 minutes obtained five minutes before obtaining liquor or abandoning the procedure.
  Rate Variability before performance Timedomain analysis: RMSDD (ms), pNN50 (%)

SECONDARY OUTCOMES:
Patients State Trait Anxiety Inventory - Short | : Five minutes before performance; Just Before Needle insertion; Five minutes after termination of the procedure
  A questionaire exploring the stress related anxiety (scores range from 6-24)
Procedure outcomes | Registered during procedure operation
  Number of needle insertions,
Procedure outcomes | Registered during procedure operation
  Failing/abandoning the procedure performance (yes/no)
Duration of time to needle insertion | Obtained during procedure, Time from needle penetration of the skin to obtaining liquor (mm:ss)
  A time stamp from first needle penetration of the skin to obtaining the liquor or abandoning the procedure.
Confidence in operator | Assessed five minutes after termination of the procedure
  A 10-point anchored Likert scale: 0=not confident - 10=very confident
Pain intensity during procedure | Assessed five minutes after termination of the procedure
  A 10-point anchored Likert scale; 0= no pain - 10= Worst imaginable pain.
Post Dural Puncture Headache | Telephone interview seven days after the procedure performance date
  Post Dural Puncture Headache, following the Lübeckers classification

CONTACTS AND LOCATIONS:
Overall Officials: Lars Konge, MD, PhD, Study Director — CAMES - Rigshospitalet
Locations (3):
- Denmark (3):
  - Department of Neurology, Rigshospitalet - Glostrup, Glostrup Municipality, Capital Region of Denmark
  - Department of Neuology, Herlev Hospital, Herlev, Capital Region of Denmark
  - Department of Neurology, University Hospital Zealand, Roskilde, Region Sjælland

IPD SHARING:
Plan to Share IPD: No